CLINICAL TRIAL: NCT06078904
Title: The Effects of Different Doses of Colchicine on High-sensitivity C-reactive Protein in Patients After Percutaneous Coronary Intervention
Brief Title: Different Doses of Colchicine on hsCRP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Xiang Cheng, Director in the department of cardiology, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: COLCRP
Record Dates: First submitted 2023-10-05; First posted 2023-10-12 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Coronary Artery Disease; Percutaneous Coronary Intervention
MeSH Terms: conditions — Coronary Artery Disease | interventions — Colchicine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Colchicine 0.5 MG (Active Comparator): Colchicine 0.5 MG, one pill a day, oral intake
  Interventions: Drug: Colchicine 0.5 MG
- Colchicine 0.375 MG (Active Comparator): Colchicine 0.375 MG, one pill a day, oral intake
  Interventions: Drug: Colchicine 0.375 MG
- Colchicine 0.25 MG (Active Comparator): Colchicine 0.25 MG, one pill a day, oral intake
  Interventions: Drug: Colchicine 0.25 MG
- Placebo (Placebo Comparator): Placebo, one pill a day, oral intake
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Colchicine 0.5 MG — Colchicine 0.5 MG, one pill a day, oral intake
  Arms: Colchicine 0.5 MG
Drug: Colchicine 0.375 MG — Colchicine 0.375 MG, one pill a day, oral intake
  Arms: Colchicine 0.375 MG
Drug: Colchicine 0.25 MG — Colchicine 0.25 MG, one pill a day, oral intake
  Arms: Colchicine 0.25 MG
Drug: Placebo — Placebo, one pill a day, oral intake
  Arms: Placebo

SUMMARY:
Colchicine reduced atherothrombotic cardiovascular events in the COLCOT and LoDoCo2 studies. US Food and Drug Administration approved colchicine as the first anti-inflammatory drug for cardiovascular diseases on June, 2023. However, there is a lack of evidence for colchicine in East Asian population with coronary heart disease, and its effectiveness and safety need further exploration. Therefore, this study aims to use different doses of colchicine to treat patients with coronary heart disease after percutaneous coronary intervention, explore the effects of different doses of colchicine on hsCRP levels, and find the optimal dose of colchicine for treating coronary heart disease in China.

ELIGIBILITY:
Inclusion Criteria:

1. Volunteer to participate, understand and sign an informed consent form;
2. Age ≥ 18 years old, regardless of gender;
3. Patient diagnosed with coronary heart disease requiring percutaneous coronary intervention;
4. Complete all planned percutaneous coronary intervention during hospitalization;
5. Patient must be treated according to national guidelines for standard treatment of coronary heart disease.

Exclusion Criteria:

1. Known allergies to colchicine;
2. Colchicine was taken within 10 days before randomization;
3. Abnormal liver function test (alanine aminotransferase >3 times the upper limit of normal value);
4. Abnormal renal function test (eGFR<30mL/min);
5. Thrombocytopenia (platelet count <100 g/L);
6. Uncontrolled infectious diseases;
7. Known immune diseases or immune-related diseases such as systemic lupus erythematosus, asthma, inflammatory bowel disease, gout, and malignant tumor, etc;
8. Pre-existing or plan for the administration of nonsteroidal anti-inflammatory drugs, hormones, immunomodulatory drugs, or chemotherapeutic drugs;
9. Pregnant women, lactating women or women of childbearing age who do not use effective contraceptives;
10. Any other circumstances in which the investigator judges that the patient is not suitable to participate in the clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2023-10-10 (Actual); Primary Completion 2023-12-25 (Actual); Study Completion 2024-04-15 (Actual)

PRIMARY OUTCOMES:
The percentage change in hsCRP | 4 weeks
  The percentage change in hsCRP compared to baseline

SECONDARY OUTCOMES:
Major adverse cardiac and cerebrovascular event (MACCE) | 4 weeks
  Composite endpoint of all cause death, non fatal myocardial infarction, non fatal stroke, and revascularization due to ischemia
Bleeding | 4 weeks
  Bleeding defined according to Bleeding Academic Research Consortium
Plasma inflammatory cytokines level | 4 weeks
  Inflammatory cytokines (IL-1β, IL-1receptor antagonist, IL-6, IL-18, tumor necrosis factor-α, myeloperoxidase, etc)
Blood drug concentrations of different doses of colchicine | 4 weeks
  Blood drug concentrations of different doses of colchicine
Expression of inflammation-related proteins in peripheral blood mononuclear cells | 4 weeks
  Inflammation-related proteins (nucleotide-binding oligomerization domain-like receptor protein 3, absent in melanoma 2, etc)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Cardiology, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fiolet ATL, Opstal TSJ, Mosterd A, Eikelboom JW, Jolly SS, Keech AC, Kelly P, Tong DC, Layland J, Nidorf SM, Thompson PL, Budgeon C, Tijssen JGP, Cornel JH. Efficacy and safety of low-dose colchicine in patients with coronary disease: a systematic review and meta-analysis of randomized trials. Eur Heart J. 2021 Jul 21;42(28):2765-2775. doi: 10.1093/eurheartj/ehab115. PMID 33769515
- [Background] Nelson K, Fuster V, Ridker PM. Low-Dose Colchicine for Secondary Prevention of Coronary Artery Disease: JACC Review Topic of the Week. J Am Coll Cardiol. 2023 Aug 15;82(7):648-660. doi: 10.1016/j.jacc.2023.05.055. PMID 37558377